CLINICAL TRIAL: NCT01203111
Title: Efficacy and Safety of Intensive Insulin Therapy With Insulin Glulisine in Patients With Type 2 Diabetes Inadequately Controlled With Basal Insulin and Oral Glucose-lowering Drugs
Brief Title: Intensive Insulin Glulisine Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Basal Insulin and Oral Glucose-lowering Drugs
Acronym: CHANGING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_R_05048; U1111-1116-3517 (Other: WHO)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine

ARMS (2):
- Intensive insulin regimen (Experimental): Treatment Period 1: Insulin glargine + metformin + other OGLDs, if any Treatment period 2: + insulin glulisine if HbA1c ≥7% at week 12 (end of treatment period 1)
  Interventions: Drug: INSULIN GLARGINE; Drug: INSULIN GLULISINE
- insulin regimen (Experimental): Treatment Period 1: Insulin glargine + metformin + other OGLDs, if any Treatment period 2: no change, if HbA1c <7% at week 12 (end of treatment period 1)
  Interventions: Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous Dose regimen: once a day in the evening at bedtime
  Other Names: Lantus SoloStar
Drug: INSULIN GLULISINE — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous Dose regimen: once a day, 0 to 15 minutes before the main meal
  Other Names: Apidra SoloStar
  Arms: Intensive insulin regimen

SUMMARY:
Primary Objective:

To evaluate the efficacy of an intensive insulin regimen with insulin glargine and insulin glulisine in terms of change in Hemoglobin A1c (HbA1c) level from week 12 (visit 7) to week 24 (visit 10).

Secondary Objectives:

1. Percentage of patients with HbA1c < 7% at week 24.
2. Percentage of patients with HbA1c < 7% and no symptomatic nocturnal hypoglycemia event at week 24.
3. Fasting Plasma Glucose (FPG) and 7-point Self Monitoring of Blood Glucose (SMBG) at week 0, week 12 and week 24.
4. Doses of insulin glargine and insulin glulisine: the daily dose (U) and the daily dose / kg (U/kg) will be calculated at week 24.
5. Systolic and diastolic blood pressure, heart rate, weight change will be measured at week 0, week 12 and week 24.
6. Number of patients suffering hypoglycemias (asymptomatic, symptomatic, nocturnal symptomatic, severe and nocturnal severe) will be evaluated during the treatment period. 7-Adverse events.

DETAILED DESCRIPTION:
The study is divided in 3 periods:

1. a 2-week run-in period,
2. a 12-week treatment period 1
3. a 12-week treatment period 2 study treatment duration per patient: 24 weeks study duration per patient: 26 weeks

ELIGIBILITY:
Inclusion criteria:

* in the run-in period:

  1. Uncontrolled Type 2 diabetes mellitus defined as HbA1c level between 7,5% and 10% assessed over the past 6 months
  2. Male or female patients from 18-75 years old inclusive
  3. Body Mass Index (BMI) between 25 and 40 kg/m2
  4. Currently treated with a basal insulin (NPH, insulin zinc or insulin detemir), plus at least 1g metformin daily, and other Oral Glucose Lowering Drug (OGLD) if any for at least 3 months
  5. Signed Informed consent obtained prior to any study procedures
* in the treatment period:

  1. HbA1c level between 7,5% and 10% assessed between week -2 and week 0
  2. Serum creatinine <= 135 µmol/L in men and <= 110 µmol/L in women
  3. Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) <= 3 times the upper limit of normal
  4. Negative pregnancy test for women of childbearing potential

Exclusion criteria:

1. Type 1 diabetes mellitus
2. Active proliferative diabetic retinopathy, defined as the application of photocoagulation or surgery performed within 6 months before study entry or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgery during the study (confirmed by an optic fundus performed over the past 2 years)
3. Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major disease making implementation of the protocol or interpretation of the study results difficult
4. History of impaired hepatic function defined as Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) greater than three times the upper limit of normal
5. History of impaired renal function defined as serum creatinine >135 µmol/l in men and > 110 µmol/l in women
6. History of drug or alcohol abuse
7. Type 2 Diabetes Mellitus (T2DM) patients treated exclusively with OGLDs
8. T2DM patients treated with an insulin other than basal insulin (Premix, rapid insulin, fast-acting insulin analogue)
9. Previous treatment with insulin glulisine
10. Concomitant treatment with thiazolidinediones, exenatide or pramlintide
11. Treatment with systemic corticosteroids within 3 months prior to study entry
12. Treatment with any investigational product within 2 months prior to study entry
13. History of hypersensitivity to the study drugs or to drugs with a similar chemical structure
14. Presence of mental condition that, in the opinion of the investigator, indicates that participation in the study is not in the best interest of the patient
15. Presence of geographic or social conditions that would restrict or limit the patient participation for the duration of the study
16. Pregnant or breast feeding women
17. Women of childbearing potential not protected by effective contraceptive method of birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c level for patients with addition of glulisine at week 12 | between week 12 and week 24 (end of treatment period)

SECONDARY OUTCOMES:
Percentage of patients with HbA1c level < 7% | at week 24 (end of treatment period)
Percentage of patients with HbA1c level < 7% and no symptomatic nocturnal hypoglycemia event | at week 24 (end of treatment period)
Fasting Plasma Glucose | at week 0, week 12 and week 24
7-point Self Monitoring of Blood Glucose | at week 0, week 12 and week 24
Daily dose of insulin glargine | at week 24 (end of treatment period)
Daily dose of insulin glulisine | at week 24 (end of treatment period)
Systolic / diastolic blood pressure, heart rate, weight change | from week 0 (baseline) to week 24 (end of treatment period)
Hypoglycemia (asymptomatic, symptomatic, nocturnal symptomatic, severe and nocturnal severe) | from week 0 (from baseline) to week 24 (end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Administrative office, Algiers, Algeria
- Administrative office, São Paulo, Brazil
- Administrative office, Netanya, Israel
- Administrative office, Beirut, Lebanon
- Administrative office, Col. Coyoacan, Mexico
- Administrative office, Casablanca, Morocco
- Administrative office, Lima, Peru
- Administrative office, Jeddah, Saudi Arabia
- Administrative office, Dubai, United Arab Emirates
- Administrative office, Caracas, Venezuela